CLINICAL TRIAL: NCT02557256
Title: Malignant Pediatric Pelvi-abdominal Tumors: A Retrospective Study
Brief Title: Malignant Pediatric Pelvic Tumors: A Retrospective Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Morsy, MD, Lecturer, Pediatric Oncology Department, Assiut University
Other Study IDs: Ped Pelvi-abd Malig
Record Dates: First submitted 2015-09-21; First posted 2015-09-23 (Estimated); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Abdominal Neoplasms; Pelvic Neoplasms
Keywords: Childhood Cancer; Abdominal Tumors; Pelvic Tumors; Pediatric Oncology
MeSH Terms: conditions — Abdominal Neoplasms; Pelvic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to retrospectively review data about malignancies that arise primarily in the pelvis and/or in the pelvic organs, in pediatric cancer patients & categorize the spectrum of these malignancies according to experience at South Egypt Cancer Institute which is the largest referral site in Upper Egypt.

DETAILED DESCRIPTION:
Background:

The newborn and infant pelvis is not fully developed and the bladder, uterus, and ovaries are to a large degree intra-abdominal. The pelvis of the infant and child has different anatomic relationships than the adolescent or adult pelvis. Neoplasms of the pediatric pelvis constitute a unique group requiring highly specialized management in a setting staffed by pediatric surgical and radiation oncologists. The most common neoplasms are rhabdomyosarcomas of the bladder, prostate, and vagina; sacrococcygeal teratoma; and the germ cell tumors, including teratomas, endodermal sinus tumors, and the choriocarcinomas. Rapidly improving chemotherapy for all of these lesions has resulted in a changed role for the surgeon.

Patients & Methods:

A hospital-based study, involving Pediatric cancer patients, those have been diagnosed with malignant tumors that primarily arising in the pelvis and/or arising from the pelvic organs, and may have an intra-abdominal extension, in the period from 2001 January till 2015 December, and received treatment at the pediatric oncology department, their medical reports will be retrospectively reviewed for data collection.

Spectrum of these malignancies will be categorized and recorded as specific disease entities, based on morphology & the primary site of occurrence, their relative incidence will be calculated, and the treatment outcomes will be verified.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose age less than 19 years.
* Patients diagnosed with a primary malignant tumor in the pelvis and/or arising from the pelvic organs.

Exclusion Criteria:

* Patients whose age more than 18 years.
* Patients diagnosed with a malignant disease primarily arising from the bone marrow.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A hospital-based study, involving Pediatric cancer patients, those diagnosed with malignant tumors of the pelvis, or arising from the pelvic organs, in the period from 2001 January till 2015 December, and received treatment at the pediatric oncology department, their medical reports will be retrospectively reviewed for data collection.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2016-01; Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Participants will be retrospectively followed forward in time from the date of initiation of treatment till the primary completion date of the study, an expected average of 5 years
  Time from the date of initiation of treatment until death from any cause.
Event Free Survival (EFS) | Participants will be retrospectively followed forward in time from the date of initiation of treatment till the primary completion date of the study, an expected average of 5 years
  Time from the date of initiation of treatment until disease progression, or death for any reason.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Groff DB. Pelvic neoplasms in children. J Surg Oncol. 2001 May;77(1):65-71. doi: 10.1002/jso.1068. PMID 11344486
- [Background] Skandalakis, J. E. and S. W. Gray (1994). Embryology for surgeons: the embryological basis for the treatment of congenital anomalies, Williams & Wilkins.